CLINICAL TRIAL: NCT03903588
Title: The Heidelberg Engineering SPECTRALIS Macular Precision and Agreement Study
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2018-2
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Retinal Layer Separation
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Normal: Eyes judged as age-appropriate normal as determined by an Investigator and that meet applicable inclusion/exclusion criteria.
  Interventions: Device: Optical Coherence Tomography
- Glaucoma: Eyes that have been diagnoses with Glaucoma
  Interventions: Device: Optical Coherence Tomography
- Retinal Disease: Eyes that have been diagnoses with a Retinal Disease
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Imaging of the Retina
  Other Names: OCT

SUMMARY:
This is a prospective clinical study that will be conducted at one clinical site located in the United States to assess two grids.

ELIGIBILITY:
Inclusion All Eye Populations

* Age 22 years or older
* Able and willing to undergo the test procedures, sign informed consent, and follow instructions
* Able to fixate
* Refraction between +6 and -6 diopters and astigmatism ≤ 2 diopters.
* Axial length ≤ 26.0 mm

Exclusion All Eye Populations

* Subjects unable to read or write
* Ocular media is not sufficiently clear to obtain acceptable quality images
* Physical inability to be properly positioned at the study devices or eye exam equipment

Inclusion Normal Population

* Eyes without prior intraocular surgery bilaterally (except cataract surgery and LASIK)
* Intraocular pressure ≤ 21mmHg
* Best corrected visual acuity ≥ 20/40
* Clinically normal appearance of the optic disc, with normal appearing neuroretinal rim with respect to color and shape, and clinically normal appearing posterior pole
* Both eyes must be determined to be normal, as determined by an investigator

Exclusion Normal Population

* Subjects with vitreal, retinal or choroidal conditions or disease of the optic nerve. Subjects may have diabetes but cannot have diabetic retinopathy.
* History of glaucoma (not including family history)
* Unreliable visual field as determined by the manufacturer's recommendations of:

Fixation losses > 20%, False Positives > 33%, False Negatives > 15%

-Visual field defects consistent with glaucomatous optic nerve damage based on at least one of the following two findings: On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level; Glaucoma hemi-field test "outside normal limits"

Inclusion Glaucoma Population

* Subjects who have a glaucoma diagnosis without prior non-glaucoma related intra-ocular surgery (except cataract surgery and LASIK)
* Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage; Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at the inferior or superior poles; or Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue

* Visual field defects consistent with glaucomatous optic nerve damage based on at least one of the following two findings:
* On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level; Glaucoma hemi-field test "outside normal limits."
* Best corrected visual acuity ≥ 20/40

Exclusion Glaucoma Population

* Subjects with presence of any ocular pathology other than Glaucoma in the study eye (cataracts are acceptable)
* Unreliable visual field as determined by the manufacturer's recommendations of:

Fixation losses > 20%, False Positives > 33%, False Negatives > 15%

Inclusion Retina Population

* Subjects who have a retinal condition diagnosis without prior non-retinal related intra-ocular surgery (except cataract surgery and LASIK).
* Intraocular pressure ≤21mmHg
* Best corrected visual acuity ≥20/400

Exclusion Retina Population

-Subjects with presence of any ocular pathology other than retinal conditions in the study eye (cataracts are acceptable)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normals, Glaucoma and Retinal Subjects as per Inclusion/Exclusion
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Retinal Layer Thickness | 5 months
  Measurement of the thickness of Retinal layers thickness to assess 2 grids

CONTACTS AND LOCATIONS:
Locations (1):
- State University of New York Optometry School, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No